CLINICAL TRIAL: NCT04985903
Title: Baby Steps III: Testing a Clinician and Patient Intervention to Promote Smoking Cessation Among Pregnant Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Pro00106131
Record Dates: First submitted 2021-07-22; First posted 2021-08-02 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-05

CONDITIONS: Smoking Cessation; Pregnancy; Communication Research
Keywords: Pregnant smokers
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: We will mask the intervention arms during the coding process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Clinicians in the intervention arm will receive a tailored communication training on smoking cessation skills and a general lecture on smoking cessation.
  Interventions: Behavioral: Clinician Communication Intervention; Other: 5A's lecture
- Control (Active Comparator): Clinicians in the control arm will be asked to attend a lecture on general information about smoking cessation for pregnant patients and smoking cessation counseling.
  Interventions: Other: 5A's lecture

INTERVENTIONS:
Behavioral: Clinician Communication Intervention — The focus of the communication program is to help clinicians increase their use of the 5 A's by improving knowledge, self-efficacy, outcome expectations, and communication skills. Training modules include didactic information with video clips of sample conversations showing specific communication skills, feedback on clinician's usage of the 5A's, and audio clips from their Pre-Intervention recorded conversations.
  Arms: Intervention
Other: 5A's lecture — a lecture on general information about smoking cessation for pregnant patients and smoking cessation counseling.

SUMMARY:
The investigators propose to conduct a combined intervention that pairs SMS smoking cessation messages for patients with individualized training for OB clinicians to improve quit rates among pregnant smoking. The aim is to determine the effect of the intervention versus control on smoking cessation outcomes on patient smoking cessation. The investigators will recruit patients at their first OB visit who report smoking at Duke and Pitt. Patients in both the control and intervention arm will receive smoking cessation support messages throughout their pregnancy. OB clinicians in the intervention arm will receive tailored smoking cessation counseling training. Clinicians in both arms will receive a one-time 5 A lecture. The investigators will analyze smoking cessation outcomes and audio recordings. This is a minimal risk study.

DETAILED DESCRIPTION:
The investigators propose a two-arm cluster randomized controlled design, in which the unit of randomization is the OB clinician. 70 OB clinicians will be randomly assigned to either the intervention or control condition. Although the unit of randomization is the clinician, the unit of evaluation is the patient: range of 6-13 patients per clinician (1-3 Pre-intervention and 5-10 Post-intervention) who receive prenatal care from enrolled OB clinicians at Duke and UPitt. The investigators will collect 3 Pre-Intervention audio-recorded initial OB visit encounters to assess pre-intervention levels of clinician communication skills and also to tailor the clinician training program. After the Pre-Intervention Phase, the investigators will randomize OB clinicians to either the intervention or control arm (see details of cluster randomization below). All OB clinicians will attend a lecture about the consequences of smoking during pregnancy and the elements of the 5 A's. Only OB clinicians randomized to the intervention arm will receive an individually-tailored, user-friendly, web-based program that teaches the 5 A's. In the Post-Intervention Phase, the investigators will assess the effect of the communication program by audio recording initial OB visits for between 5-10 pregnant women who smoke for each OB clinician in both arms (n=542 total). The investigators will provide all patients the SMS text-delivered intervention. Additionally, the investigators will survey these patients before their visit, immediately after their visit, at the end-of-pregnancy, and 6-weeks postpartum. Due to anticipated study attrition, the investigators will recruit up 80 clinicians and 700 patients at both sites until the investigators reach a complete data set for our desired sample size. Biochemically validated smoking cessation at end-of-pregnancy is the primary outcome (Aim 1). To assess Aim 2, investigators will code for clinician use of the 5 A's in the audio-recorded encounters and analyze patient perceptions of the communication from post-encounter data and the post-study survey for clinicians. To assess Aim 3, investigators will collect smoking status at 6 weeks postpartum.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Receiving prenatal care from an enrolled OB clinician
* Self-report smoking tobacco at their first OB visit
* Access to a cell phone with texting capabilities

Exclusion Criteria:

* Unable to speak and read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2022-03-25 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Number of Patients in the Post-Intervention Phase With Validated Cessation | End-of-pregnancy, up to 45 minutes
  Biochemically validated (urine cotinine) 7-day point prevalent as defined by urine cotinine levels below 50ng/ML.

SECONDARY OUTCOMES:
Number of A's performed in the Post-Intervention Phase for each Clinician | Post-intervention recordings (all recording will happen prior to giving birth), up to 12 weeks
  Obtained by coding 11 recordings of patient encounters in the Post-Intervention Phase. We will follow a codebook to assess the number of A's performed in the Post-Intervention visits for each clinician. Coders will also assess whether each Advice segment is clear, strong, or personalized. We will assign advice a score of 0-3 with a score of 3 indicating highest quality of advice.
Mean rated autonomy support for each Post-intervention patient | Baseline, up to 15 minutes
  6-item Health care climate questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn I Pollak, PhD, Principal Investigator — Duke University
Locations (1):
- Durham OB, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No